CLINICAL TRIAL: NCT06518590
Title: Effect of Single-versus Double-limb Cycling Exercise on Blood Flow in Patients With Peripheral Artery Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Merna Marwan Mohamed Kamal, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cyling on blood flow in PAD
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group(A) (Active Comparator): Twenty five patients will receive unilateral limb training sequentially (counter weighted single limb cycling ) (dominant limb, then non-dominant limb) by bicycle for 20-30 minutes per session, three sessions per week for 2 months (8 weeks), in addition to health advices and their medications
  Interventions: Device: Cycle
- Group(B) (Active Comparator): Twenty-five patients will receive bilateral limbs training by bicycle for 20_ 30 minutes per session, three sessions per week for 2 months (8 weeks), in addition to health advices and their medications
  Interventions: Device: Cycle
- Group(C) (Active Comparator): Twenty five patients will receive medications in addition to health advices.
  Interventions: Device: Cycle

INTERVENTIONS:
Device: Cycle — Kettler upright bike Giro P:

SUMMARY:
This study will be conducted to investigate the effect of single limb cycling exercise and the effect of double limb cycling exercise on blood flow in patients with peripheral artery disease and compare between both effects.

DETAILED DESCRIPTION:
Global populations are undergoing a major epidemiological transition in which the burden of atherosclerotic cardiovascular diseases is shifting rapidly from high-income to low-income and middle-income countries (LMICs). Peripheral artery disease (PAD) is no exception, so that greater focus is now required on the prevention and management of this disease in less-advantaged countries (Gerry et al., 2017) PAD prevalence and incidence are both sharply age-related, rising >10% among patients in their 60s and 70s. With the aging of the global population, it seems likely that PAD will be increasingly common in the future. Prevalence seems to be higher among men than women for more severe or symptomatic disease (Michael et al., 2015).

PAD causes leg pain, impaired health-related quality of life, immobility, tissue loss and a high risk of major adverse events, including myocardial infarction, stroke, revascularization, amputation and death. The drug cilostazol, exercise therapy and revascularization are the current treatment options for the limb symptoms of PAD, but each has limitations (Jonathan et al., 2022) Few studies conducted the importance of active and passive movements and aerobic exercises for Cardiovascular especially peripheral artery disease patients as mentioned previously, thus the aim of this study is to conduct single limb cycling exercise and double limbs cycling exercise to PAD patient to determine the effect of cycling on blood flow velocity and which is more effective and leads to more benefits compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* 1. Mild to moderate PAD ( ABI ranges from less than 0.90 to 0.50) 2. Intermittent claudication / Typical claudication 3. Their age will be ranged from 50_60 years old. 4. Quitting smoking for more than 3 months 5. Body mass index (BMI) from 25.0 to 29.9kg/m2.

Exclusion Criteria:

* 1. Patients with uncontrolled pulmonary disease. 2. Patients with vascular severe complication as critical limb ischemia(ABI less than 0.5) 3. Patients with unstable angina, uncontrolled cardiac arrhythmia, decompensated heart failure.

  5. Patients with severe musculoskeletal problems (e.g., severe knee osteoarthritis or post knee replacement surgeries).

  6. Any patients who missed more than two weeks of the program or want to terminate the program.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Blood flow velocity by Doppler | baseline
  Blood flow (velocity) and circulation: which will be measured by the doppler ultrasonogrophy at the begining and at the end of the study.
  - Doppler ultrasonogrophy of the lower extremity arteries, from common femoral to pedal arteries peak systolic velocity (PSV) recorded in meters per second (Ugwu.,et al .,2021 ) .The normal peak systolic velocity (PSV ) in peripheral lower limb arteries varies from 45-180 cm/s .
  Severe arterial disease manifests as a PSV in excess of 200 cm/s , monophasic waveform and spectral broading of the doppler wave form .

SECONDARY OUTCOMES:
Functional capacity test (6 Min walk test ) | baseline
  Functional capacity which will be : measured by a Six min walk test before and after the program of exercising according to the American Thoracic Society 113, TECHNICAL ASPECTS OF THE 6MWT (at the beginning and at the end of the study).
The ankle -brachial index test | baseline
  which will be measured by Duplex at the beginning and at the end of the program of exercising
Walking impairment questionnaire | baseline
  Walking impairment questionnaire: An effective tool to assess the effect of treatment in patients with intermittent claudication.
  WIQ is a valid tool to detect improvement or deterioration in the daily walking ability of patients with intermittent claudication.

REFERENCES:
- [Background] Firnhaber JM, Powell CS. Lower Extremity Peripheral Artery Disease: Diagnosis and Treatment. Am Fam Physician. 2019 Mar 15;99(6):362-369. PMID 30874413
- [Background] Bevan GH, White Solaru KT. Evidence-Based Medical Management of Peripheral Artery Disease. Arterioscler Thromb Vasc Biol. 2020 Mar;40(3):541-553. doi: 10.1161/ATVBAHA.119.312142. Epub 2020 Jan 30. PMID 31996023